CLINICAL TRIAL: NCT00836264
Title: Pharmacogenomic Analysis of Morphine Pharmacokinetics and Response Variability Following Pediatric Tonsillectomy and Adenoidectomy: A Genome-Wide Association Approach
Brief Title: Pharmacogenomics Analysis of Morphine Pharmacokinetics in Pediatric Tonsillectomy and Adenoidectomy
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: 08-007023
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Tonsillectomy; Adenoidectomy; Pharmacokinetics
Keywords: Morphine; Phenotype; Genotype; Tonsillectomy; Adenoidectomy; Opioid Receptors; Genome-Wide Association; Pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — PK plasma samples will be obtained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Morphine T & A: Subjects ages 4-18 years of age who have a Tonsillectomy and Adenoidectomy and receive morphine for pain control and who have also enrolled in the CAG study at CHOP, "A Study of the Genetic Causes of Complex Pediatric Disorders" (GCPD study), as approved by the CHOP IRB, 2006-7-4886.

SUMMARY:
Intravenous (IV) morphine requirement for immediate postoperative pain control depends upon the complex interplay of patient history, wound severity, environment, and genetics. Even for relatively uniform stimulus intensity, such as that associated with tonsillectomy and adenoidectomy (T&A), there can be marked individual variability in response to morphine. Some patients are refractory to standard doses and need increased amounts. Others are sensitive, require less drug to attain acceptable pain levels, and/or experience unwanted side effects that limit dosing. A significant number must be switched to different analgesics altogether. Despite the long clinical history of morphine as a postoperative analgesic, researchers have only begun to examine the origins of response variability.

The investigators will look at 2000 retrospective Tonsillectomy and Adenoidectomy (T&A) cases and using this data and incorporating additional patient, surgical, and environmental factors that may contribute to response variability, the investigators then propose a prospective genome-wide association (GWA) study of 1500 children ages 4 to 18 years treated with IV morphine sulfate for day surgery T&A.

DETAILED DESCRIPTION:
Morphine Tonsilectomy and Adenoidectomy (T&A) Pharmacokinetics (PK) study will be done as a part of the larger institutional Center for Applied Genomics (CAG) project entitled "A Study of the Genetic Causes of Complex Pediatric Disorders" (GCPD study), as approved by the Children's Hospital of Philadelphia (CHOP) IRB, 2006-7-4886. By combining Genome Wide Association (GWA) and PK data, we wish to conduct a Pharmacogenomic (PG) study of IV morphine administered as standard of care during and after pediatric day surgery T&A. Because we expect several genes to play a role in the morphine response, we must use a large, relatively uniform pediatric surgical population such that for T&A. Through observation and minimal-risk blood sampling of this cohort of children, we hope to identify genetic variants that predict analgesic response to (and serum levels of) morphine sulfate. Pediatric patients ages 4-18 y, presenting with significant tonsillar/adenoidal tissue hypertrophy, sleep disordered breathing and/or recurrent infection, and requiring T&A are eligible. Morphine is the most common IV analgesic used for T&A at the Children's Hospital of Philadelphia (CHOP). As is necessary for accurately defining analgesic response phenotype, morphine will be administered in a structured manner consistent with standard of care at this institution. As defined below, children resistant to morphine (MR) and those sensitive to it (MS) will be identified as specific phenotypes to be compared with normal responders (NR) in a GWA study.

This study begins with a retrospective electronic database query of 2000 day surgery T&A cases between 11/1/2005 and 10/31/2008 in which morphine was used as the sole IV analgesic. Data from this portion of the study will help us refine phenotype parameters, should robust subpopulations of response types emerge, and provide background information required for eventual project funding by the National Institutes of Health (NIH). The prospective portion of the study will follow an additional 1650 children newly enrolled in the CAG study and now presenting for T&A.

ELIGIBILITY:
Inclusion Criteria:

1. Concurrent enrollment in the GCPD study (IRB 2006-7-4886)
2. Scheduled for day surgery T&A with expected same day discharge at CHOP Main in Philadelphia, Pennsylvania (PA) or the CHOP Ambulatory Surgical Facilities (ASFs) in Chalfont, PA; Exton, PA; or Voorhees, New Jersey (NJ)
3. Male or female, age 4 - 18 years, all races and ethnic backgrounds
4. Able to self-report pain on the Faces Pain Scale - Revised (FPS-R).
5. Informed consent as addendum to GCPD consent document
6. Assent for children ≥7 years of age

Exclusion Criteria:

1. Parents/guardians or subjects who, in the opinion of the investigator, may be non-compliant with study schedules or procedures
2. Non-English speaking subjects or parents. The reliability of the morphine analgesic requirement phenotype could be adversely affected by subtle communication differences between subjects and nursing staff assessing pain and administering morphine during patient recovery should language barriers exist. Parents must also be fluent in English as they will be at the bedside shortly after their child's arrival in recovery and could influence how their child understands pain scoring and how they interact with the nursing and research staff.
3. Those parents/guardian or subjects not consenting to, or willing to participate in the GCPD study (IRB 2006-7-4886).
4. Patients < 4 y of age were excluded to improve phenotype reliability. Due to a higher empirical risk of postoperative obstruction following T&A, children < 4 years of age are admitted for overnight observation. The titration of morphine is more difficult in these patients as clinicians generally follow more restrictive dosing regimens and the total morphine dose is drawn out over an extended period. Furthermore, the self-report Faces Pain Scale - Revised (FPS-R) has been validated for children ≥ 4 y and will be used to corroborate the morphine response phenotypes that are primarily based on morphine doses administered to achieve low Face, Legs, Activity, Cry, Consolability (FLACC) scores. The latter behavioral scoring is required for early morphine administration as children and adolescents emerging from anesthesia may have difficulty expressing themselves in the first 30 min. In addition, it is important for the study statistical analysis to have a sequential scoring system over time that is applicable to all ages. Finally, the incidence of emergence agitation/delirium, a clinical phenomenon that shares some features of pain, but becomes distinct over 15-30 minutes, is higher in younger patients. (Sikich, 2004; Vlajkovic, 2007) By excluding children < 4 years Investigators decrease the proportion of subjects whose FLACC scores may be high on the basis of emergence agitation/delirium.
5. Significant comorbid conditions requiring a non-standard anesthetic regimen such as a history of severe post-operative nausea and vomiting requiring propofol infusion, a total intravenous anesthestic (TIVA) technique and/or mandating planned post-operative hospital admission.
6. Documented allergy or adverse reaction to morphine in the patient.
7. Use of opioids (e.g. codeine, oxycodone, morphine, hydromorphone) within the previous month.
8. Use of non-steroidal anti-inflammatory agents or acetaminophen in the 3 days preceding the T&A. No acetaminophen will be included in the premedication regimen on the day of surgery.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children having Tonsillectomy and Adenoidectomy procedures done at The Children's Hospital of Philadelphia, at the Main Hospital and also at the satellite surgical centers, who have also consented to participate in "A Study of the Genetic Causes of Complex Pediatric Disorders" (GCPD study), as approved by the CHOP IRB, 2006-7-4886.
Sampling Method: Non-Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be to identify genetic variants that contribute to the variability of morphine analgesic response following pediatric day surgery T&A. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Cook-Sather, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States